CLINICAL TRIAL: NCT03694392
Title: Examining Vaccine Effectiveness (VE) of Flublok Relative to Standard Dose Inactivated Influenza Vaccine Among Kaiser Permanente Northern California Members Aged 18-64 Years
Brief Title: Flublok v. Standard Dose Vaccine Effectiveness Among Kaiser Permanente Northern California Adults 18-64 Years
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CN-18-3176
Record Dates: First submitted 2018-09-27; First posted 2018-10-03 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Influenza; Pneumonia; Lower Respiratory Tract Infection; Acute Myocardial Infarction; Congestive Heart Failure; Stroke
Keywords: influenza; vaccine effectiveness
MeSH Terms: conditions — Influenza, Human; Pneumonia; Heart Failure; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flublok Recipients: Kaiser Permanente Northern California members aged 18-64 years who receive Flublok Quadrivalent vaccine.
  Interventions: Biological: Flublok Quadrivalent
- SD-IIV Recipients: Kaiser Permanente Northern California members aged 18-64 years who receive standard dose inactivated influenza vaccine (SD-IIV).
  Interventions: Biological: Standard Dose Inactivated Influenza Vaccine (SD-IIV)

INTERVENTIONS:
Biological: Flublok Quadrivalent — Flublok Quadrivalent vaccine is a recombinant hemagglutinin influenza vaccine indicated for active immunization against disease caused by influenza A subtype viruses and type B viruses contained in the vaccine for adults 18 years of age and older. Use of recombinant DNA techniques to produce vaccine antigen expressed in cell culture is a method that avoids growing the influenza viruses in embryonated hen's eggs.
  Groups: Flublok Recipients
Biological: Standard Dose Inactivated Influenza Vaccine (SD-IIV) — For the 2018-2019, 2019-2020, and 2020-2021 flu seasons, the primary SD-IIVs used will be Fluarix Quadrivalent and Flulaval Quadrivalent.
  Groups: SD-IIV Recipients

SUMMARY:
The overall objective of this study is to describe the effectiveness of Flublok Quadrivalent vaccine compared to standard dose inactivated influenza vaccine (SD-IIV) in adults 18 through 64 years of age. During this study, Flublok Quadrivalent or SD-IIV will be administered according to the guidelines in the Prescribing Information materials and only to persons for whom it is indicated. The 2018-2019, 2019-2020, and 2020-2021 formulations of recombinant influenza vaccine (Flublok Quadrivalent vaccine) and SD-IIV will be evaluated for outcomes including all polymerase chain reaction (PCR)-confirmed influenza, PCR-confirmed hospitalized influenza, hospitalized community-acquired pneumonia and cardio-respiratory events.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of ≥18 and <65 years at the time of influenza vaccination
* Receive either Flublok Quadrivalent vaccine or standard dose inactivated influenza vaccine at a Kaiser Permanente Northern California facility during the study period from August 2018 through April 2020

Exclusion Criteria:

* Children <18 years old
* Adults ≥65 years old

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligible adults aged 18-64 years will receive either Flublok Quadrivalent vaccine or a standard dose inactivated influenza vaccine in the course of routine influenza vaccination during each of the two influenza seasons of the study period at Kaiser Permanente Northern California.
Sampling Method: Probability Sample
Enrollment: 2776278 (Actual)
Dates: Start 2018-09-16 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola P Klein, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California (entire region), Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No
All data reported to Sanofi Pasteur by the Kaiser Permanente Northern California Vaccine Study Center will be deidentified and aggregated.

REFERENCES:
- [Derived] Hsiao A, Yee A, Izikson R, Fireman B, Hansen J, Lewis N, Gandhi-Banga S, Selmani A, Talanova O, Kabler H, Inamdar A, Klein NP. Safety of quadrivalent recombinant influenza vaccine in pregnant persons and their infants. AJOG Glob Rep. 2024 Sep 20;4(4):100395. doi: 10.1016/j.xagr.2024.100395. eCollection 2024 Nov. PMID 39512761
- [Derived] Hsiao A, Yee A, Fireman B, Hansen J, Lewis N, Klein NP. Recombinant or Standard-Dose Influenza Vaccine in Adults under 65 Years of Age. N Engl J Med. 2023 Dec 14;389(24):2245-2255. doi: 10.1056/NEJMoa2302099. PMID 38091531
- [Derived] Hsiao A, Hansen J, Nunley KV, Lewis N, Selmani A, Inamdar A, Mallett-Moore T, Izikson R, Rudin D, Klein NP. Safety of recombinant quadrivalent influenza vaccine compared to inactivated influenza vaccine in Chinese adults: An observational study. Vaccine. 2022 Jan 31;40(5):774-779. doi: 10.1016/j.vaccine.2021.12.035. Epub 2022 Jan 6. PMID 34998605

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flublok Recipients | SD-IIV Recipients
Started | 1018043 | 1758235
Completed | 632962 ("Completed" refers to final analysis study population (as opposed to reflecting drop-out, etc.). All individuals included at the start were vaccinated as part of routine clinical care. "Not Completed" refers to vaccinated individuals who were not included in the final analysis due to not being part of the randomization process or other reasons.) | 997366 ("Completed" refers to final analysis study population (as opposed to reflecting drop-out, etc.). All individuals included at the start were vaccinated as part of routine clinical care. "Not Completed" refers to vaccinated individuals who were not included in the final analysis due to not being part of the randomization process or other reasons.)
Not Completed | 385081 | 760869

BASELINE CHARACTERISTICS:
Population: Final analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | Flublok Recipients | SD-IIV Recipients | Total
Number analyzed (Participants) | 632962 | 997366 | 1630328
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 632962 | 997366 | 1630328
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363921 | 585482 | 949403
  Male | 269041 | 411884 | 680925
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 275117 | 420570 | 695687
  Black | 27601 | 45674 | 73275
  Asian | 159104 | 255008 | 414112
  Pacific Islander | 4824 | 7499 | 12323
  Native American | 2908 | 4635 | 7543
  Multiracial | 16229 | 25946 | 42175
  Unknown/Other | 147179 | 238034 | 385213
Region of Enrollment [Number; unit: participants]
  United States | 632962 | 997366 | 1630328
History of asthma [Count of Participants; unit: Participants] | 86127 | 132550 | 218677
History of diabetes [Count of Participants; unit: Participants] | 67026 | 97192 | 164218
History of chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 6174 | 8563 | 14737
History of coronary heart disease [Count of Participants; unit: Participants] | 11947 | 16902 | 28849
Receipt of influenza vaccine in previous year [Count of Participants; unit: Participants] | 414500 | 640263 | 1054763
Charlson Comorbidity Index [Count of Participants; unit: Participants]
  No Charlson comorbidities | 508118 | 812879 | 1320997
  CCI=1 | 81980 | 122562 | 204542
  CCI≥2 | 42864 | 61925 | 104789
Body mass index [Count of Participants; unit: Participants]
  0 - < 18.5 kg/m² | 7819 | 12311 | 20130
  18.5 - < 25 kg/m² | 188431 | 306194 | 494625
  25 - < 30 kg/m² | 206663 | 323624 | 530287
  ≥ 30 kg/m² | 209817 | 321607 | 531424
  None | 20232 | 33630 | 53862
Number of weeks with outpatient visits in prior year [Count of Participants; unit: Participants]
  0 | 57602 | 92349 | 149951
  1-3 | 270701 | 427043 | 697744
  4-7 | 165444 | 256965 | 422409
  ≥8 | 139215 | 221009 | 360224
Number of inpatient stays in prior year [Count of Participants; unit: Participants]
  0 | 573712 | 902365 | 1476077
  1 | 44860 | 71208 | 116068
  2 | 9707 | 15896 | 25603
  3 | 2885 | 4735 | 7620
  ≥4 | 1798 | 3162 | 4960
Prior membership [Count of Participants; unit: Participants]
  <1 year | 78004 | 127160 | 205164
  1 to <2 years | 62407 | 100315 | 162722
  2 to <3 years | 52678 | 84938 | 137616
  3 to <4 years | 45919 | 74028 | 119947
  4 to <5 years | 41545 | 66292 | 107837
  ≥5 years | 352409 | 544633 | 897042

OUTCOME MEASURES:

1. Primary Outcome: Number of Adults 50-64 Years Old With Polymerase-chain Reaction (PCR) Confirmed Influenza Tests
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed for whether they had a PCR-confirmed positive influenza test (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30).
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
participants | 559 | 925
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox — Adjustment for multiplicity for the secondary outcomes was performed with the use of Holm's adjustment method; Models were adjusted for age, age squared, sex, and race or ethnic group after weighting with stabilized facility-specific propensity scores; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.76 to 0.94] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 15.3% (5.9%, 23.8%)

2. Secondary Outcome: Number of Adults 50-64 Years Old Hospitalized With PCR-confirmed Influenza
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed for whether they had an inpatient stay and had a PCR-confirmed positive influenza test (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30).
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
participants | 95 | 153
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox — Adjustment for multiplicity for the secondary outcomes was performed with the use of Holm's adjustment method; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.65 to 1.09] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 15.9% (-9.2% to 35.2%)

3. Secondary Outcome: Number of Adults 50-64 Years Old Hospitalized With Community-acquired Pneumonia
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed for whether they had an inpatient stay for community-acquired pneumonia (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30).
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
Participants | 106 | 183
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox — Adjustment for multiplicity for the secondary outcomes was performed with the use of Holm's adjustment method; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.66 to 1.06] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 16.7% (-5.6% to 34.4%)

4. Secondary Outcome: Number of Adults 50-64 Years Old Hospitalized With Cardio-respiratory Events
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed for whether they had an inpatient stay for cardio-respiratory events (e.g., pneumonia, other lower respiratory infections, acute myocardial infarction, congestive heart failure, stroke) (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30).
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
Participants | 631 | 890
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox — Adjustment for multiplicity for the secondary outcomes was performed with the use of Holm's adjustment method; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.88 to 1.08] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 2.4% (-8.1% to 11.9%)

5. Other Pre Specified Outcome: Number of Adults 18-49 Years Old Hospitalized With Community-acquired Pneumonia
Description: as for outcome 3
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
Participants | 37 | 49
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.75 to 1.80] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: -15.7% (-79.5% to 25.5%)

6. Other Pre Specified Outcome: Number of Adults 50-64 Years Old With Influenza-Like Illness (ILI)
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30) for influenza-like illness (ILI) International Classification of Diseases, 10th Edition (and absence of a negative lab-confirmed influenza)
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
Participants | 1826 | 2871
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.001, 95% CI 2-sided [0.95 to 1.06] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: -0.1% (-6.0% to 5.4%)

7. Other Pre Specified Outcome: Number of Adults 50-64 Years Old With All-Cause-Hospitalizations
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30) for all-cause hospitalizations
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
Participants | 4308 | 6005
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.8, 95% CI 2-sided [-2.2 to 5.5] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 1.8% (-2.2% to 5.5%)

8. Other Pre Specified Outcome: Number of Adults 50-64 Years Old With All-Cause Mortality
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30) for all-cause mortality
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
Participants | 286 | 422
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 9.4, 95% CI 2-sided [-5.4 to 22.1] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 9.4% (-5.4% to 22.1%)

9. Other Pre Specified Outcome: Number of Adults 18-49 Years Old With Polymerase-chain Reaction (PCR) Confirmed Influenza Tests
Description: as for outcome 1
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
participants | 827 | 1510
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.86 to 1.02] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 6.2% (-2.2% to 13.9%)

10. Other Pre Specified Outcome: Number of Adults 18-49 Years Old Hospitalized With PCR-confirmed Influenza
Description: as for outcome 2
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
participants | 48 | 88
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.75 to 1.52] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: -6.9% (-51.6% to 24.6%)

11. Other Pre Specified Outcome: Number of Adults 18-49 Years Old Hospitalized With Cardio-respiratory Events
Description: as for outcome 4
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
Participants | 133 | 208
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.76 to 1.12] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 5.2% (-18.8% to 24.4%)

12. Other Pre Specified Outcome: Number of Adults 18-49 Years Old With Influenza-Like Illness (ILI)
Description: as for outcome 6
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
Participants | 2904 | 5434
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.85 to 0.93] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 10.8% (6.6% to 14.7%)

13. Other Pre Specified Outcome: Number of Adults 18-49 Years Old With All-Cause-Hospitalizations
Description: as for outcome 7
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
Participants | 1858 | 2950
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.001, 95% CI 2-sided [0.94 to 1.06] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: -0.1% (-6.2% to 5.6%)

14. Other Pre Specified Outcome: Number of Adults 18-49 Years Old With All-Cause Mortality
Description: as for outcome 8
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
Participants | 66 | 79
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [1.06 to 2.00] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: -45.5% (-100.2% to -5.8%)

15. Other Pre Specified Outcome: Number of Adults 18-49 Years Old With Polymerase-chain Reaction (PCR) Confirmed Influenza A Tests
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed for whether they had a PCR-confirmed positive influenza A test (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30).
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
participants | 682 | 1282
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.82 to 0.99] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 10.2% (1.4% to 18.2%)

16. Other Pre Specified Outcome: Number of Adults 18-49 Years Old With Polymerase-chain Reaction (PCR) Confirmed Influenza B Tests
Description: Patients who receive either Flublok or SD-IIV will be retroactively assessed for whether they had a PCR-confirmed positive influenza B test (≥14 days after vaccination) as recorded in their electronic medical record by the end of the influenza season (April 30).
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 353562 | 601514
participants | 146 | 231
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.95 to 1.43] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: -16.2% (-43.0% to 5.5%)

17. Secondary Outcome: Number of Adults 50-64 Years Old With Polymerase-chain Reaction (PCR) Confirmed Influenza A Tests
Description: as for outcome 15
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
participants | 522 | 862
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.76 to 0.94] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 15.7% (6.0% to 24.5%)

18. Secondary Outcome: Number of Adults 50-64 Years Old With Polymerase-chain Reaction (PCR) Confirmed Influenza B Tests
Description: as for outcome 16
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Flublok Recipients | SD-IIV Recipients
Number analyzed (Participants) | 279400 | 395852
participants | 37 | 64
Statistical Analysis 1: Comparison: Flublok Recipients vs SD-IIV Recipients; Test type: Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.60 to 1.34] — Relative vaccine effectiveness (95% CI) calculated as 1 minus the hazard ratio, expressed as a percentage: 10.3% (-33.9% to 39.9%)

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | Flublok Recipients | SD-IIV Recipients
All-Cause Mortality (participants affected / at risk) | 352/632962 | 501/997366
Serious Adverse Events (participants affected / at risk) | 0/632962 | 0/997366
Other Adverse Events (participants affected / at risk) | 0/632962 | 0/997366

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03694392/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03694392/SAP_001.pdf